CLINICAL TRIAL: NCT06933030
Title: Assessment of Customized 3D Zirconium Versus Titanium Mesh for Anterior Maxillary Ridge Augmentation With Delayed Implant Placement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Mostafa Alhashash, ASSISTANT LECTURER, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMPDR7-242235
Record Dates: First submitted 2025-03-06; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Ridge Augmentaton and Dental Implants; Bone Loss, Alveolar
Keywords: ridge augmentation; dental implant; titanium mesh; zirconium mesh
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: Group I (controlled group):
  - Ten sites of anterior maxillary ridge atrophy will be treated by titanium mesh with bone graft with delayed implant placement.
  Group II (tested group):
  - Ten sites anterior maxillary ridge atrophy will be treated by zirconium mesh with bone graft with delayed implant placement.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (controlled group): - (Other): Group I (controlled group):
  - Ten sites of anterior maxillary ridge atrophy will be treated by titanium mesh with bone graft with delayed implant placement.
  Interventions: Device: titanium mesh with bone graft with delayed implant placement.
- Group II (tested group): (Experimental): Group II (tested group):
  - Ten sites anterior maxillary ridge atrophy will be treated by zirconium mesh with bone graft with delayed implant placement.
  Interventions: Device: zirconium mesh with bone graft with delayed implant placement.

INTERVENTIONS:
Device: titanium mesh with bone graft with delayed implant placement. — titanium mesh with bone graft with delayed implant placement.
  Arms: Group I (controlled group): -
Device: zirconium mesh with bone graft with delayed implant placement. — zirconium mesh with bone graft with delayed implant placement.
  Arms: Group II (tested group):

SUMMARY:
The aim of the present study is to assess the customized 3D zirconium versus titanium mesh for anterior maxillary ridge augmentation with delayed implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Patients from both genders with the age range of 18-60 years with good systemic health, no contraindication for periodontal surgery and able to maintain good oral hygiene.
  2. Patient with anterior maxillary alveolar ridge deficiency (horizontal, vertical or combined defects) less than 2 mm in width or less than 6 mm in height - measured from the alveolar crest to the basal bone in order to be enrolled in this study. (56)
  3. Adequate zone of keratinized gingiva at minimum 3mms.
  4. Patient with sufficient inter-arch space for future dental rehabilitation.
  5. Subjects who are not on any medication known to interfere with periodontal tissue health or healing within 6 months of the study.

Exclusion Criteria:

Exclusion Criteria:

1. History of systemic diseases (i.e. diabetes, autoimmune dysfunction, prolonged cortisone therapy, or chemotherapy) that would contraindicate periodontal surgical treatment or affect bone turn over.
2. Patients with deleterious habits like the use of tobacco chewing or smoking ones.
3. History of previous periodontal surgical treatment of the involved sites.
4. Presence of malocclusion and pathologic movement of teeth in involved sites.
5. Patient not willing to give consent for the study and poor plaque control.(57)
6. Pregnant or nursing mothers.
7. Patients with acute odontogenic infection.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation | 6 months
  The patients will be followed up clinically postoperatively every 48-72 hours for the first week then after 2weeks then one month and then after 3 months then after 6 months for preserving: Presence/absence of mesh instability, flap dehiscence, exposed mesh, bone graft loss outside the flap, hematoma or laceration.

SECONDARY OUTCOMES:
radiographic bone volume | 6,12 months
  A CBCT will be done preoperatively (base line) and after 6 months and finally after 12 months postoperatively to assess dimensions of newly formed bone and its density.
histologically | 6 months
  The bone cores, left inside the trephine burs will be carefully rinsed with a cold 5% glucose solution. The specimens will be fixed in 10% formalin solution at pH 7.2 for a week and dehydrated with a graded series of alcohols. After the pre-infiltration treatment the bone cores will then be completely embedded in 100% resin until the specimens became transparent. Finally, the bone cores will be oriented and polymerized.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt